CLINICAL TRIAL: NCT05125666
Title: Efficacy of Dual Task Training on Children With Ataxia After Medulloblastoma Resection: (A Randomized Controlled Trial)
Brief Title: Efficacy of Dual Task Training on Children With Ataxia After Medulloblastoma Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Mostafa Sedeek Selim, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTT-Ataxia-1
Record Dates: First submitted 2021-10-02; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Ataxia; Medulloblastoma
MeSH Terms: conditions — Ataxia; Medulloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Task Training (Experimental)
  Interventions: Other: Dual Task Training (Motor + Cognitive)
- Ordinary Physical Therapy for Ataxia (Active Comparator)
  Interventions: Other: Traditional Regular Exercise

INTERVENTIONS:
Other: Dual Task Training (Motor + Cognitive) — Each child in this group will perform one-hour session consist of two tasks (cognitive and balance task) in addition to the traditional physical therapy program three times weekly for 8 successive weeks.
  Arms: Dual Task Training
Other: Traditional Regular Exercise — Each child in this group will receive the selected physical therapy program which include mobility exercises, strengthening exercises, balance exercises, gait training exercises, and exercises to improve physical conditioning for one-hour session three times weekly for 8 successive weeks.
  Arms: Ordinary Physical Therapy for Ataxia

SUMMARY:
The aim of this study is to evaluate the effect of using a selected dual-task- training program to improve postural stability in children with ataxia after medulloblastoma resection. Thirty patients will participate in this study. Patients will be classified randomly into two equal groups: study and control groups -Both groups will receive conventional physical therapy treatment including mobility exercises, balance exercises, gait training exercises, and exercises to improve physical conditioning. In addition, the study group will receive a selected dual-task training program including balance and cognitive activities. The treatment program will be conducted three days per week for eight successive weeks. The patients will be assessed with the Scale of Assessment and Rating of Ataxia, Humac Balance System, the Pediatric Balance Scale and Functional Independent Measurement. The measures will be recorded two times: before the application of the treatment program (pre) and after the end of the treatment program (post).

ELIGIBILITY:
Inclusion Criteria:

All children with the following criteria will be in rolled in the study

1. Age range from (5-10 years).
2. Severity of ataxia will be from 15-30 by SARA scale.
3. Children after 2 months of medulloblastoma resection.
4. They can stand and walk with minimal support.
5. They have good cognition, compliance, and ability to understand and instructions.
6. Children receiving radiotherapy and chemotherapy sessions
7. They are medically stable

Exclusion Criteria:

Children will be excluded from the study if they have

1. Any neuromuscular disorder.
2. Visual impairment.
3. Cognitive problem
4. Convulsion.
5. Peripheral neuropathy due to chemotherapy.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Static balance of patients with ataxia after resection measured by center of pressure using force plate mode in the humac balance system. | 2 months
Improvement in dynamic balance of patients with ataxia after resection measured by using tilt mode in the humac balance system. | 2 months
Improvement in Activities of Daily Living (ADL) measured by functional independence measurement. | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- 57357 Children Cancer Hospital, Cairo, El Sayeda Zainab, Egypt

IPD SHARING:
Plan to Share IPD: No